CLINICAL TRIAL: NCT03212677
Title: Safe and Effective Delivery of Supplemental Iron to Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Simin Meydani, Vice Provost for Research; Director, Nutritional Immunology Lab, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPP1139998
Record Dates: First submitted 2017-06-22; First posted 2017-07-11 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2021-04

CONDITIONS: Iron
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Iron-deficient children (Active Comparator): Previously iron-deficient children aged 6-24 months on iron therapy. Ferrous sulfate administered at 4 mg Fe/kg/d per standard of care.
  Interventions: Dietary Supplement: Ferrous sulfate
- Non-iron-deficient children (No Intervention): Non-iron-deficient children aged 6-24 months used as a reference.
- Adult Placebo (Placebo Comparator): Iron-replete postmenopausal women, and men, receiving placebo daily for 4 weeks.
  Interventions: Other: Placebo
- Adult Ferrous sulfate daily (Experimental): Iron-replete postmenopausal women, and men, receiving ferrous sulfate daily (containing 60 mg Fe per day) for 4 weeks. In Phase II, iron-replete postmenopausal women, and men, receiving ferrous sulfate daily (containing 120 mg Fe per day) for 4 weeks.
  Interventions: Dietary Supplement: Ferrous sulfate
- Adult ferrous sulfate weekly (Experimental): Iron-replete postmenopausal women, and men, receiving ferrous sulfate weekly (containing 60 mg Fe per day) for 4 weeks.
  Interventions: Dietary Supplement: Ferrous sulfate
- Adult ferrous sulfate + micronutrient (Experimental): Iron-replete postmenopausal women, and men, receiving ferrous sulfate + micronutrient supplement (containing 60 mg Fe per day) for 4 weeks.
  Interventions: Dietary Supplement: Ferrous sulfate
- Adult IHAT (Experimental): Iron-replete postmenopausal women, and men, receiving IHAT (containing 60 mg Fe per day) for 4 weeks. In Phase II, iron-replete postmenopausal women, and men, receiving IHAT (containing 120 mg Fe per day) for 4 weeks
  Interventions: Dietary Supplement: IHAT
- Adult Aspiron (Experimental): Iron-replete postmenopausal women, and men, receiving Aspiron (containing 60 mg Fe per day) for 4 weeks. In Phase II, iron-replete postmenopausal women, and men, receiving Aspiron (containing 120 mg Fe per day) for 4 weeks.
  Interventions: Dietary Supplement: Aspiron

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — Standard-of-care therapy for iron deficiency anaemia
  Arms: Adult Ferrous sulfate daily; Adult ferrous sulfate + micronutrient; Adult ferrous sulfate weekly; Iron-deficient children
Dietary Supplement: IHAT — IHAT is a nanoparticle composed of three General Regarded As Safe (GRAS) substances, iron hydroxide, tartaric acid and adipic acid. The particle itself resembles the normal metabolite ferritin, which is a larger polyatomic particle. Like ferritin, IHAT can be absorbed by endocytosis, but dissociates within the enterocyte and is subsequently metabolized as ferrous iron.
  Other Names: Iron hydroxide adipate tartrate
  Arms: Adult IHAT
Dietary Supplement: Aspiron — Aspiron is a product of the natural fermentation of Koji (Aspergillus oryzae) in the presence of ferrous sulfate. The iron-rich koji biomass is heated, harvested and dried which results in the inactivation of Koji powder that contains 8-10% iron. Koji (A. oryzae) is widely used for making such foods as soy sauce, tempeh, miso, and for producing food-grade α-amylase, and is considered safe by Joint Food and Agriculture Organization of the United Nations (FAO)/WHO Committee on Food Additives and has been accepted as a GRAS constituent of food.
  Other Names: Aspiron™ Natural Koji Iron
  Arms: Adult Aspiron
Other: Placebo — Cornstarch
  Other Names: Melogel Cornstarch
  Arms: Adult Placebo

SUMMARY:
Iron deficiency-related anemia is the most common nutritional deficiency disorder in the world, mainly affecting children, women and older adults in underdeveloped countries. To combat iron deficiency, inorganic forms of iron (such as ferrous sulfate) are often used as an iron supplement. One big problem is that high levels of this kind of iron supplement produce negative health effects. This includes diarrhea, changes in the bacteria in the gut, as well as increased severity to malaria in young children in countries with high rates of that parasite.

Most forms of iron are not well absorbed and, therefore, pass through the intestine to be eliminated in the stool. This unabsorbed iron can be used by gut bacteria, disturbing the balance of healthful and potentially harmful bacteria in the colon, which can increase inflammation in the body.

In this study, the investigators are seeking to determine whether two new forms of iron cause fewer changes in the gut bacteria thus lowering inflammation while providing similar amounts of iron to the body. The findings from this research study are important because they will inform the development of safer treatments for iron deficiency.

DETAILED DESCRIPTION:
The forms of iron currently available have serious adverse effects that limit their use in addressing prevalent iron deficiency. Iron-supplementation programs have been frustrated by the serious side effects of inorganic forms of iron, which, due to low enteric absorptive efficiency, must be given in relatively high levels (5-20 fold effective levels of heme-iron in foods). Those adverse effects include infectious diarrhea, changes in the gut microbiome and increased serious morbidity among iron-replete children in malaria-endemic areas. The underlying causes of these effects are thought to involve stress on the gut due to excess unabsorbed iron, which can be pro-oxidative and pro-inflammatory. In addition, unabsorbed, soluble iron can be used by the gut microbiome and favor the proliferation of pathogenic enteric bacteria which can contribute to the inflammatory response that leads to down-regulation of iron absorption. Lack of a safe and effective treatment leaves large numbers of children iron deficient, many with associated anemia. Thus, the burden of disease, which includes growth, cognitive and physical performance deficits as well as increased risk of infection, continues to climb in this age group.

The overall goal of this project is to generate evidence to support development of a modality of providing bioavailable iron that does not or produces less adverse effects in iron-replete individuals. The investigators will employ the commonly used iron supplement FeSO4 to compare with two novel forms of iron with features that suggest each may be a useful nutritional source of iron with fewer side effects than FeSO4. The first novel form of iron is a nanoparticulate formulation of iron hydroxide adipate tartrate (IHAT). The second novel form of iron is an organic fungal iron metabolite, Aspiron, which has recently been developed by using a food-grade Aspergillus oryzae cultured in iron-fortified media.

The investigators will evaluate these forms of iron using a randomized clinical trial approach that will robustly test the formal hypotheses and yield useful answers to the primary questions about the relative safety and efficacy of these novel forms of iron in iron-replete subjects. This study is divided to two phases. In Phase I, the investigators will determine of effects of form of low-dose, supplemental iron. Three forms of iron administered at the dose of 60 mg Fe/d will be evaluated against the primary outcomes of ex vivo malarial infectivity, bacterial proliferation potential (also assessed ex vivo) and gut inflammation, and other relevant outcomes in adults. In this protocol the investigators refer to this set of indicators as the "safety profile". The justification for providing 60 mg Fe/d is based on the World Health Organization (WHO) recommendation for daily supplementation for non-anemic, pregnant women with 30-60 mg Fe/d. In addition, the effects on those outcomes of ferrous sulfate administered daily (60 mg Fe/d) vs. weekly (420 mg Fe administered in one weekly dose) will be compared. There is great practical value in addressing this hypothesis of whether a weekly dose can be administered without adverse effects. Nested within this design will be a second comparative study of effects in iron-replete children and adults to validate the applicability of data obtained in adults to children.

For the forms of iron found to produce no adverse effects at the 60 mg Fe/d dose level, Phase II of the study will be conducted in which such forms will be tested at a higher, therapeutic dose of 120 mg Fe/d against the same outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 50-80 years
* BMI range: 18-35
* Men and post-menopausal women (defined as no menses for > 1year or S/P hysterectomy with bilateral oopherectomy)
* Typical bowel pattern: at least 1 stool every other day
* Willing to take iron and be randomized into study intervention group
* Willing to abstain from recreational drug use and consumption > 2 alcoholic drinks per day during study participation
* Will not be undergoing colonoscopy in the 2 months before, or during the course of the study

Exclusion Criteria:

* Any major illness or condition that may interfere with study outcomes at the discretion of the study MD
* Personal history of G-6-P (glucose-6-phosphate dehydrogenase) deficiency
* Diabetes Type 1 & Type 2 or use of any pharmacological treatment for diabetes
* Endocrine disorders including diabetes, unstable thyroid disease (dose adjustment of thyroid replacement in the past 6 months), adrenal disease, pheochromocytoma or parathyroid disease
* Recent history of inflammatory diseases (for example: rheumatoid arthritis, lupus)
* Use tumor necrosis factor (TNF) blockade medication, methotrexate, or other immune-modulating drugs
* Steroid use (except for non-prescription topical and nasal steroids, e.g. Flonase)
* If participant is on hormone replacement therapy with estrogen, testosterone or growth hormone, has the dosage regimen changed in the past month, or expected to change during course of study
* History of myocardial infarction, stroke or transient ischemic attack (TIA), coronary artery bypass graft, stenosis >50% diagnosed within the past 1 year or acute unstable cardiovascular disease.
* Clotting/bleeding disorders or ongoing anticoagulant use: coumadin (warfarin), Eliquis, Xarelto, Pradaxa
* GI diseases, conditions or medications known to influence GI absorption including active peptic ulcer disease or inflammatory bowel disease (such as ulcerative colitis, Crohn's disease), pancreatic insufficiency, celiac disease, malabsorption disorders (other than lactose intolerance)
* Hx of stomach or bowel resection (other than appendectomy), gastric bypass or other bariatric weight loss procedure
* Regular use (> 2 times per week) of acid lowering medication: antacids, proton pump inhibitors (PPI), H2 blockers
* History of eating disorder anorexia, bulimia or binge-eating in the past 5 years
* Actively undergoing dialysis
* Inadequately controlled hypertension (HTN) @ the discretion of study MD or Registered Nurse
* Certain psychiatric disorders including schizophrenia, bipolar major depression or psychosis (depression OK, if stable on treatment regimen for > 6 months)
* Immunodeficiency condition, HIV or AIDS
* Cancer of any type (except for non-melanoma skin) in past year
* Actively using cancer chemotherapeutic agents
* Regular use of acetylsalicylic acid (ASA); NSAIDs; Cox-2 inhibitors. However, infrequent NSAID use (not on a regular scheduled basis) allowed if able to hold NSAIDs x 72 hours prior to all blood draws
* Infection or febrile illness within 2wks prior to study or study blood draws, may rescheduled >2wks after resolution of symptoms
* Hx of malaria; or vaccination or treatment for malaria, or antimalarial prophylaxis in past 3 months
* Seizure disorders (OK if well managed with medication: no seizure activity x 3 yrs)
* Hx splenectomy
* Chronic liver disease such as hepatitis B, C or cirrhosis
* Use of fiber supplements, laxatives or stool softeners, unless willing to maintain consistent dose for 2 weeks prior to entry and for duration of study
* Colonoscopy procedure or prep within 2 months prior to or during study
* Antibiotic use (including dental prophylaxis use within 3 months prior to or during study participation). Non-prescription topical antibiotics OK.
* If using probiotic or prebiotic foodstuffs or pills/capsules, will dosage regimen change during course of study?
* Inability to deliver stool sample to center within 18 hours of bowel movement
* Alcohol use on average > 2 servings/day or > 14 servings/wk (Serving size: 12oz beer/4oz wine/2oz hard liquor) or self-reported binge drinking
* Current use of iron supplement or other nutritional supplements containing iron
* Use of dietary supplements containing vitamins (except Ca+, Vit D), minerals, herbal other plant-based preparations, fish oil supplements (including cod liver oil) or homeopathic remedies x 2 weeks prior to or during study. If individual wishes to participate, must stop these supplements >2 weeks prior to study.
* Inadequate venous access or history of a bilateral mastectomy with nodal dissection
* Participation in other research study during the same time period
* No social security number (required for stipend payment)
* Iron saturation outside of normal range
* Hemoglobin (Hgb) < 11.7 (females) < 13.2 (males)
* Serum creatinine > 1.5 mg/dl
* Fasting blood sugar >126 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) > 1.5x upper range of normal
* Serum glutamic-pyruvic transaminase (SGPT) > 1.5x upper range of normal mg/dl in absence of benign cause, i.e.: Gilbert's syndrome

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Malaria infectivity | 4 weeks
  Malaria (Plasmodium falciparum) infectivity of host erythrocytes will be assessed in vitro
Bacterial proliferation potential | 4 weeks
  Bacterial proliferation potential studies will be conducted in vitro using subject plasma
Fecal calprotectin | 4 weeks
  Fecal calprotectin will be analyzed using ELISA.

SECONDARY OUTCOMES:
Biochemical markers of systemic inflammation, such as plasma cytokines | 4 weeks
Biochemical markers of intestinal inflammation, such as fecal cytokines | 4 weeks
Intestinal microbiome | 4 weeks
Fecal short chain fatty acids | 4 weeks
Biochemical markers of redox stress, such as F2α-isoprostanes | 4 weeks
Biochemical markers of iron status, such as ferritin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simin N Meydani, DVM, PhD, Principal Investigator — Tufts Univeristy; Gerald F Combs, PhD, Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lewis ED, Ortega EF, Dao MC, Barger K, Mason JB, Leong JM, Osburne MS, Magoun L, Nepveux V FJ, Chishti AH, Schwake C, Quynh A, Gilhooly CH, Petty G, Guo W, Matuszek G, Pereira D, Reddy M, Wang J, Wu D, Meydani SN, Combs GF Jr. Safe and effective delivery of supplemental iron to healthy adults: a two-phase, randomized, double-blind trial - the safe iron study. Front Nutr. 2023 Oct 11;10:1230061. doi: 10.3389/fnut.2023.1230061. eCollection 2023. PMID 37899826
- [Derived] Lewis ED, Wu D, Mason JB, Chishti AH, Leong JM, Barger K, Meydani SN, Combs GF. Safe and effective delivery of supplemental iron to healthy older adults: The double-blind, randomized, placebo-controlled trial protocol of the Safe Iron Study. Gates Open Res. 2021 Feb 9;3:1510. doi: 10.12688/gatesopenres.13039.2. eCollection 2019. PMID 33655197